CLINICAL TRIAL: NCT02234050
Title: Trabectedin for Recurrent Grade II or III Meningioma: a Randomized Phase II Study of the EORTC Brain Tumor Group
Brief Title: Trabectedin for Recurrent Grade II/III Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1320-BTG; 2014-002446-47 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-09-09 (Estimated); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Recurrent High Grade Meningioma
Keywords: Grade 2 Chordoid meningioma; Grade 2 Clear cell meningioma; Grade 2 Atypical meningioma; Grade 3 Papillary meningioma; Grade 3 Rhabdoid meningioma; Grade 3 Anaplastic meningioma; Grade 3 Malignant meningioma
MeSH Terms: interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trabectedin (Experimental): Patient will be treated with trabectedin
  Interventions: Drug: Trabectedin
- Local standard of care (Other): Treatment in the control arm is left to the discretion of the investigator, according to the local standard of care.
  Interventions: Other: Local standard of care

INTERVENTIONS:
Drug: Trabectedin — Trabectedin will be given as a 24-hour infusion every 3 weeks at a starting dose of 1.5 mg/m2 body surface area (BSA), until one of the treatment withdrawal criteria has been met.
  Other Names: Yondelis
  Arms: Trabectedin
Other: Local standard of care — Left to the discretion of the investigator
  Arms: Local standard of care

SUMMARY:
The aim of this study is to collect data on activity, toxicity and quality of life of trabectedin therapy in patients with recurrent high-grade meningioma.

DETAILED DESCRIPTION:
This is a randomized open label multicenter comparative phase II trial. The objective of the study is to investigate whether trabectedin demonstrates sufficient antitumor activity against recurrent grade II or III to justify further investigation in phase III or as adjuvant therapy for newly diagnosed disease after resection and radiotherapy.

ELIGIBILITY:
Patient selection criteria

* Age 18 or older
* Histological diagnosis of World Health Organization (WHO) grade II (chordoid meningioma, clear cell meningioma, atypical meningioma) or WHO grade III (papillary meningioma, rhabdoid meningioma, anaplastic/malignant meningioma) according to WHO 2007 classification.
* Radiologically documented progression of any existing tumor (growth > 25% in the last year) or appearance of new lesions (including intra- and extracranial manifestations)
* No more option for local therapy (resection or radiotherapy) after maximal feasible surgery and radiotherapy
* No prior systemic anti-neoplastic therapy for meningioma
* Measurable disease (10 x10 mm) on cranial MRI no more than 2 weeks prior to randomization.
* WHO performance status 0-2
* Adequate liver, renal and hematological function within 4 weeks prior to randomization, defined as:

  * Neutrophils ≥ 1.5 x 109/L, hemoglobin ≥ 9 g/dL or hemoglobin ≥ 5.6 mmol/L, platelets ≥ 100 x 109/L
  * Total Bilirubin ≤ 1 x Upper Limit of Normal (ULN), serum glutamate pyruvate transaminase(SGPT)/ Alanine Aminotransferase (ALT) and serum glutamate oxaloacetate transaminase (SGOT)/ Aspartate Aminotransferase (AST) ≤ 2.5 x ULN
  * Alkaline phosphatase ≤ 2.5 x ULN; if alkaline phosphatase > 2.5 ULN, Alkaline Phosphatase (ALP) hepatic isoenzyme and/or 5-nucleotidase and/or gamma glutamyltransferase (GGT) must be within the normal range
  * Albumin ≥ 30 g/L
  * Serum creatinine ≤ 1.5 x ULN
  * Creatinine clearance > 30 ml/min as calculated by Cockcroft and Gault formula (see Appendix E)
  * Creatine phosphokinase (CPK) ≤ 2.5 x ULN
* Normal cardiac function (LVEF assessed by Multigated radionuclide angiography (MUGA) or Echocardiogram (ECHO) within normal range of the institution), normal 12 lead ECG (without clinically significant abnormalities). The following unstable cardiac conditions are not allowed:

  * Congestive heart failure
  * Angina pectoris
  * Myocardial infarction within 1 year before registration/randomization
  * Uncontrolled arterial hypertension defined as blood pressure ≥ 150/100 mm Hg despite optimal medical therapy
  * Arrhythmias clinically significant
* Life expectancy of at least 9 weeks
* No history of any other invasive malignancy within the last 5 years (except adequately treated non-melanoma skin cancer, clinically localized and very low risk prostate cancer, and adequately treated cervical intraepithelial neoplasia)
* No serious illness or medical conditions, specifically: active infectious process; chronic active liver disease, including chronic hepatitis B, C or cirrhosis
* No concomitant use of any other investigational agent or phenytoin
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to the first dose of study treatment. Women of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 3 months after the last study treatment. Men who are fertile must use effective contraception during treatment with trabectedin and for 5 months thereafter. A highly effective method of birth control is defined as one that results in low failure rate, i.e. less than 1% per year, when used consistently and correctly.
* Female subjects who are breastfeeding should discontinue nursing prior to the first dose of study treatment and until 3 months after the last study treatment.
* No known MRI or CT, including contrast media, contraindications
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Patients with a buffer range from the normal values of +/- 5 % for hematology and +/- 10% for biochemistry are acceptable. A maximum of +/- 2 days for timelines may be acceptable
* Before patient randomization, written informed consent must be given according to International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH)/ Good Clinical Practice (GCP), and national/local regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07 (Actual); Study Completion 2019-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Preusser, Study Chair — Medical University Vienna - General Hospital AKH
Locations (47):
- Austria (2):
  - Landesnervenklinik Wagner Jauregg, Linz
  - Medical University Vienna - General Hospital AKH, Vienna
- Belgium (5):
  - Hopitaux Universitaires Bordet-Erasme - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - CHU Dinant Godinne - UCL Namur, Yvoir
- France (10):
  - CHU de Bordeaux - Groupe Hospitalier Saint-André - Hopital Saint-Andre, Bordeaux
  - CHU de Lyon - CHU Lyon - Hopital neurologique Pierre Wertheimer, Bron
  - Centre Georges-Francois-Leclerc, Dijon
  - CHRU de Lille, Lille
  - Centre Leon Berard, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - CHU de Nice - Hopital Pasteur, Nice
  - Assistance Publique - Hopitaux de Paris - La Pitie Salpetriere, Paris
  - Centre Eugene Marquis, Rennes
  - Gustave Roussy, Villejuif
- Germany (10):
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum - Essen, Essen
  - Klinikum Der J.W. Goethe Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg - Klinik fuer Neurochirurgie, Freiburg im Breisgau
  - Universitaetsklinikum Heidelberg - UniversitaetsKlinikum Heidelberg - Head Hospital, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Ludwig-Maximilians-Universitaet Muenchen - Klinikum der Universitaet Muenchen - Campus Grosshadern, München
  - Universitaetsklinikum Muenster, Zentralklinikum, Münster
  - Universitaetskliniken Regensburg, Regensburg
  - Eberhard Karls Universitaet Tuebingen - Universitaetsklinikum Tuebingen, Tübingen
- Italy (5):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Ospedale San Raffaele, Milan
  - Istituto Oncologico Veneto IRCCS - Ospedale Busonera, Padua
  - Istituto Regina Elena / Istituti Fisioterapici Ospitalieri, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino - Ospedale San Giovanni - Dipartimento Neuroscienze, Torino
- Netherlands (3):
  - Spaarne Gasthuis - Vrije Universiteit Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus MC Cancer Institute - location Daniel den Hoed, Rotterdam
- Oslo University Hospital - Radiumhospitalet, Oslo, Norway
- Spain (5):
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Barcelona
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), L'Hospitalet de Llobregat
  - Hospital Universitario 12 De Octubre, Madrid
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (4):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol
  - NHS Lothian - Western General Hospital, Edinburgh
  - Guy's and St Thomas' NHS - St Thomas Hospital, London
  - Newcastle Hospitals NHS Trust - Freeman Hospital, Northern Centre For Cancer Care, Newcastle

REFERENCES:
- [Derived] Hundsberger T, Surbeck W, Hader C, Putora PM, Conen K, Roelcke U. [Meningioma: management of the most common brain tumour]. Praxis (Bern 1994). 2016 Apr 13;105(8):445-51. doi: 10.1024/1661-8157/a002320. German. PMID 27078728

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient randomization was only accepted from authorized investigators. Patients were randomized directly on the EORTC online randomization system (ORTA = online randomized trials access), accessible 24 hours a day, 7 days a week, through the internet. A patient could only be randomized after verification of eligibility. Both the eligibility check and randomization Case Report Forms had to be done before the start of the protocol treatment.
Groups:
- Local Standard of Care: Treatment in the control arm is left to the discretion of the investigator, according to the local standard of care.
  Local standard of care: Left to the discretion of the investigator. In some countries no treatment is administered to the patient instead an active surveillance or wait and see approach is applied. This was also considered a valid local standard of care in this study.
Period: Overall Study
Arm/Group | Trabectedin | Local Standard of Care
Started | 61 | 29
Completed | 0 | 4
Not Completed | 61 | 25
Not completed — Lack of Efficacy | 38 | 22
Not completed — Adverse Event | 13 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Sponsor's decision | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Standard of Care | Trabectedin | Total
Number analyzed (Participants) | 29 | 61 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 29 | 45
  >=65 years | 13 | 32 | 45
Age, Continuous [Median (Full Range); unit: years] | 63 [38.9 to 81.3] | 62 [21.2 to 80.1] | 62.2 [21.2 to 81.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 31 | 43
  Male | 17 | 30 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 61 | 90
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 5 | 6
  Netherlands | 2 | 3 | 5
  Belgium | 1 | 5 | 6
  Norway | 2 | 2 | 4
  Italy | 5 | 14 | 19
  United Kingdom | 5 | 7 | 12
  France | 9 | 14 | 23
  Germany | 2 | 5 | 7
  Spain | 2 | 6 | 8
World Health Organization (WHO) performance status [Number; unit: participants] — The WHO performance status (PS) classification is used to assess the functional status of patients, PS 0: Fully active, able to carry on all activities without restriction. PS 1: Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work PS 2: Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours. PS 3: Capable of only limited self-care; confined to bed or chair more than 50% of waking hours. Lower scores for better outcomes. Higher scores for poorer outcomes.
  participants
    PS 0 | 7 | 15 | 22
    PS 1 | 13 | 34 | 47
    PS 2 | 9 | 11 | 20
    PS 3 | 0 | 1 | 1
Histology grade [Number; unit: participants] — The World Health Organization (WHO) meningioma grading system classifies into grades based on their histopathological characteristics. WHO Grade II (Atypical) : these meningiomas are considered atypical and have a higher likelihood of recurrence compared to Grade I (benign). WHO Grade III (Anaplastic/Malignant): these are the least common but most aggressive type of meningiomas. They have the highest risk of recurrence and can metastasize. The grading system helps in guiding the treatment approach and predicting the prognosis of individuals with meningiomas.
  participants
    WHO Grade II | 19 | 36 | 55
    WHO Grade III | 10 | 25 | 35
Corticosteroids intake [Number; unit: participants]
  No | 20 | 39 | 59
  Yes | 9 | 21 | 30
  Not completed | 0 | 1 | 1
Largest diameter of initial target lesions (mm) [Median (Full Range); unit: mm] | 36 [13 to 115] | 44 [14 to 86] | 43.5 [13 to 115]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression (PD) was measured according to the Macdonald response criteria as at least a 25% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) AND an absolute increase of ≥ 5 mm. Appearance of new lesions will also constitute PD (including lesions in previously unassessed areas). Progression Free Survival (PFS) was measured from the date of randomization until the date of first objective progression or the date of patient's death whichever occurs first. Patients without evidence of progression was censored at the last follow-up visit date. If a patient received a second anti-tumoral therapy without prior documentation of disease progression, the patient was censored at the date of starting new anti-tumoral therapy.
Time Frame: From the date of randomization until the date of first objective progression or the date of patient's death whichever occurs first up.PFS was assessed by its median the point time at which 50% of the patients have experienced disease progression or death.
Population: Per protocol population was defined as all patients who were eligible and had started their allocated treatment (at least one dose of Trabectedin or start of local standard of care therapy)
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Trabectedin: Patient will be treated with trabectedin Trabectedin: Trabectedin will be given as a 24-hour infusion every 3 weeks at a starting dose of 1.5 mg/m2 body surface area (BSA), until one of the treatment withdrawal criteria has been met.
Arm/Group | Local Standard of Care | Trabectedin
Number analyzed (Participants) | 22 | 57
Months | 4.17 [2.00 to 5.95] | 2.43 [2.07 to 3.32]
Statistical Analysis 1: Comparison: Local Standard of Care vs Trabectedin; Test type: Superiority; p = 0.204, Regression, Cox; Hazard Ratio (HR) = 1.42, 80% CI 2-sided [0.997 to 2.028]

2. Secondary Outcome: Progression Free Survival at 6 Months (PFS-6)
Description: The PFS probability at 6 months (PFS-6) was extracted from the Kaplan-Meyer PFS curve. 95% confidence intervals were computed based on the Greenwood's formula.
Time Frame: From the date of randomization until the date of first objective progression or the date of patient's death whichever occurs first. PFS at 6 months,the proportion of patients who have not experienced disease progression or death by 6 months is presented
Population: Per protocol population: all patients who were eligible and had started their allocated treatment (at least one dose of Trabectedin or start of local standard of care therapy)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Local Standard of Care | Trabectedin
Number analyzed (Participants) | 22 | 57
percentage of participants | 29.1 [11.9 to 48.8] | 21.1 [11.3 to 32.9]

3. Secondary Outcome: Objective Response (CR/PR)
Description: Tumor response was measured according to the Macdonald response criteria as Complete Response (CR): disappearance of all target and non-target lesions. Residual lesions (other than nodes < 10 mm) thought to be non-malignant should be further investigated before CR can be accepted. Clinical evaluation must be stable or improving. No steroids should be needed.
  Partial Response (PR): at least a 50% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the baseline sum of diameters. Non target lesions must be non-PD. Clinical evaluation must be stable or improving. Steroid dose must be stable or diminishing. Objective response was defined as both CR and PR. It was scheduled every 9 weeks from randomization until progression and after discontinuation of treatment without progression, every 9 weeks for the first year from randomization and every 12 weeks thereafter.
Time Frame: From the date of randomization until disease progression or death, up to 24 months from date of randomization.It was assessed every 9 or 12 weeks (see measure description for details).The response rate presented is based on the best response observed.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Local Standard of Care | Trabectedin
Number analyzed (Participants) | 22 | 57
percentage of participants | 0 | 1.8

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was calculated from the date of randomization up to the date of death (any cause). For patients still alive or lost to follow-up at the time of analysis, survival will be censored at last follow-up visit date.
Time Frame: From the date of randomization up to the date of death. OS was assessed by its median the point time at which 50% of the patients have experienced death.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Local Standard of Care | Trabectedin
Number analyzed (Participants) | 22 | 57
Months | 10.61 [5.91 to 13.54] | 11.37 [8.15 to 16.89]
Statistical Analysis 1: Comparison: Local Standard of Care vs Trabectedin; Test type: Superiority; p = 0.94, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.53 to 1.71]

5. Secondary Outcome: Health-related Quality of Life (HRQol)
Description: Due to the small sample size and low compliance in the Standard of Care (SoC) arm, the analysis of Quality of Life (QoL) was restricted to describing The Global health status / QoL scores at baseline. The Global health status / QoL scores are part of the EORTC QLQ-C30, which is a core questionnaire designed to assess the quality of life of cancer patients. These scores are derived from a specific scale within the EORTC Quality of Life Questionnaire (QLQ-C30) that evaluates the overall health status and quality of life of the patient. The scoring for the Global health status / QoL scale involves a linear transformation of the raw score to a standardized score ranging from 0 to 100. This scale is revised in version 3.0 of the QLQ-C30 and includes two items with a range of 6, specifically items 29 (Global health status)and 30 (QoL scale). Higher score values represent a better outcome i.e. a higher quality of life.
Time Frame: Baseline measurements were collected before or on the day of the start of protocol treatment, but no earlier than 28 days before. The median baseline Global health status / QoL scores per treatment arm is reported.
Population: Safety population: all patients who had started their allocated treatment (at least one dose of Trabectedin or start of local standard of care therapy). Additionally per protocol windows were used to allocate the Qol assessments to the baseline timepoint.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Local Standard of Care | Trabectedin
Number analyzed (Participants) | 24 | 55
score on a scale | 54.2 [16.7 to 83.3] | 58.3 [0 to 100]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of treatment (Trabectedin or SOC) up to 27 months after patient enrolment in the study. All-Cause Mortality was assessed through study completion, up to 36 months after patient enrolment in the study.
Description: Both serious and non-serious AEs were collected. We reported serious adverse events (SAEs) and all AEs. Non serious AEs are accounted for in the all AEs report. All AEs report is included in the Other (Not Including Serious) section. SAEs and all AEs were reported in the safety population defined as the randomized patients who have started their allocated treatments. All-cause mortality was also reported in the safety population.
Arm/Group | Trabectedin | Local Standard of Care
All-Cause Mortality (participants affected / at risk) | 40/61 | 17/27
Serious Adverse Events (participants affected / at risk) | 26/61 | 4/27
Other Adverse Events (participants affected / at risk) | 58/61 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=61) | Local Standard of Care (N=27)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Other AE (Blood and lymphatic system disorders) | 3 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Other AE (Ear and labyrinth disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Other AE (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Sudden Death Nos (General disorders) | 1 | 0
Other AE (Hepatobiliary disorders) | 3 | 0
Catheter Related Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Mucosal Infection (Infections and infestations) | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Wound Infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Cpk Increased (Investigations) | 1 | 0
Ggt Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracranial Hemorrhage (Nervous system disorders) | 2 | 0
Ischemia Cerebrovascular (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Other AE (Nervous system disorders) | 0 | 1
Other AE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=61) | Local Standard of Care (N=27)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Other AE (Blood and lymphatic system disorders) | 3 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Vestibular Disorder (Ear and labyrinth disorders) | 1 | 0
Other AE (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Blurred Vision (Eye disorders) | 1 | 0
Eyelid Function Disorder (Eye disorders) | 0 | 1
Watering Eyes (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 15 | 3
Diarrhea (Gastrointestinal disorders) | 9 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Esophageal Pain (Gastrointestinal disorders) | 0 | 1
Fecal Incontinence (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 2 | 0
Mucositis Oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 29 | 5
Periodontal Disease (Gastrointestinal disorders) | 0 | 1
Stomach Pain (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 22 | 3
Other AE (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Edema Limbs (General disorders) | 3 | 1
Fatigue (General disorders) | 26 | 11
Fever (General disorders) | 6 | 2
Flu Like Symptoms (General disorders) | 1 | 2
Gait Disturbance (General disorders) | 4 | 0
Localized Edema (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 2 | 1
Sudden Death Nos (General disorders) | 1 | 0
Other AE (Hepatobiliary disorders) | 5 | 0
Bladder Infection (Infections and infestations) | 1 | 1
Bronchial Infection (Infections and infestations) | 0 | 1
Catheter Related Infection (Infections and infestations) | 3 | 0
Device Related Infection (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 1
Eye Infection (Infections and infestations) | 1 | 1
Gum Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Mucosal Infection (Infections and infestations) | 1 | 1
Otitis Externa (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Skin Infection (Infections and infestations) | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 2
Wound Infection (Infections and infestations) | 1 | 1
Other AE (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Cpk Increased (Investigations) | 1 | 0
Ggt Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 3 | 1
Serum Amylase Increased (Investigations) | 1 | 0
Weight Gain (Investigations) | 6 | 0
Weight Loss (Investigations) | 9 | 3
White Blood Cell Decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 11 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Other AE (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Weakness Right-Sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Other AE (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 2 | 0
Cerebrospinal Fluid Leakage (Nervous system disorders) | 1 | 0
Cognitive Disturbance (Nervous system disorders) | 2 | 1
Concentration Impairment (Nervous system disorders) | 0 | 1
Depressed Level Of Consciousness (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 3 | 2
Dysgeusia (Nervous system disorders) | 2 | 2
Dysphasia (Nervous system disorders) | 2 | 1
Edema Cerebral (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 10 | 7
Hydrocephalus (Nervous system disorders) | 2 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Intracranial Hemorrhage (Nervous system disorders) | 3 | 0
Ischemia Cerebrovascular (Nervous system disorders) | 0 | 2
Ivth Nerve Disorder (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 2
Paresthesia (Nervous system disorders) | 3 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 2
Pyramidal Tract Syndrome (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 6 | 4
Somnolence (Nervous system disorders) | 2 | 0
Stroke (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 1
Trigeminal Nerve Disorder (Nervous system disorders) | 1 | 0
Other AE (Nervous system disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 4 | 2
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Other AE (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 3 | 0
Genital Edema (Reproductive system and breast disorders) | 1 | 0
Testicular Disorder (Reproductive system and breast disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Other AE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 2
Other AE (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 9 | 11
Hypotension (Vascular disorders) | 3 | 0
Thromboembolic Event (Vascular disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT02234050/Prot_SAP_000.pdf